CLINICAL TRIAL: NCT06419153
Title: Evaluating the Efficacy of the Sub-psoas Fascial Plane Block for Post-operative Analgesia Following Hemiarthroplasty
Status: Not yet recruiting | Type: Observational
Sponsor: University College Hospital Galway (Other)
Collaborators: Prof John McDonnell (Unknown); Prof John Laffey (Unknown)
Responsible Party: Principal Investigator, Orla Murphy, Dr Orla Murphy, Specialist Registrar Anaesthesia, University College Hospital Galway
Other Study IDs: C.A. 3190
Record Dates: First submitted 2024-05-04; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Hemiarthroplasty
Keywords: anaesthesia, regional; SPF block; hemiarthroplasty; subpsoas fascia block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SPF Block Group: In this RCT, all patients enrolled will be undergoing Emergency HemiArthroplasty in the theatre complex in University Hospital Galway.
  Under ultrasound-guidance the SPF will be performed by the experienced consultant anaesthesiologist, whereby 30ml of 0.75% Ropivicaine will be slowly injected into the subpsoas fascial plane, whilst at all times throughout and following the procedures the patient will be closely haemodynamically monitored. The patient will be followed up in the recovery post-anaesthetic care unit up to four hours following their surgery. They will then be reviewed by the one of the co-investigators at a timeframe of 0-24 hours and 24-48 hours post-operatively to further establish their analgesic efficacy, their pain scores (see supplementary appendix), quality of recovery, time to remobilization and opioids requirements, ensuring the patient is comfortable and aiming to maximize their recovery period.
- No SPF Block Group: In this RCT, all patients enrolled will be undergoing Emergency HemiArthroplasty in the theatre complex in University Hospital Galway
  Participants randomized to 'standard care' will receive the standard care required as determined by the treating team in the form of intravenous analgesia.

SUMMARY:
The study aims to examine the efficacy and safety of an ultrasound-guided regional anaesthetic technique intended to provide pain relief following hip surgery. It involves targeting a layer of tissue known as the psoas fascia, where the nerves of the lumbar plexus, supplying the lower limb, are located. There are many well-established ultrasound-guided techniques that target similar anatomical planes and structures, such as the psoas compartment block and quadratus lumborum plane block, which are widely used in clinical practice. This is not a new technique but rather a new approach to a well-established and utilized technique (the psoas compartment block). Early remobilisation plays a key role in the recovery of post-operative patients, helping to reduce the incidence of pneumonia, deep vein thrombosis, and delirium. By reducing motor weakness while still providing adequate pain relief and minimizing the use of strong painkillers such as morphine, it will help to reduce the risk of falls and length of hospital stay. An initial case series in GUH has previously followed a small cohort of patients who, following informed consent, underwent the subpsoas fascia plane (SPF) block vs. suprainguinal fascia iliaca block as part of their multimodal pain relief following surgery. It was found that in this group there was a reduction in postoperative pain scores, decreased use of strong painkillers, and earlier time to remobilisation.

DETAILED DESCRIPTION:
Background:

Hip fracture surgery is one of the commonest orthopaedic operations performed in the Republic of Ireland, and is associated with significant patient morbidity, mortality and health care costs. The National Irish Hip Fracture Report recorded 1,950 hip fractures in 2013, 71% were female and the highest proportions were in the 80-89 age group. It has been estimated that the overall prevalence of hip fractures is projected to increase in line with increasing elderly population and projected demographic changes.

Early remobilization has become a key integral component of the optimal post-surgical management of hip fractures. Based on the National Institute for Health and Care Excellence (NICE) guidance, the National Hip Fracture UK Database has adopted patient remobilisation on the day of or day after surgery as a key performance indicator. Early mobilisation has been shown to reduce the risk of in-hospital mortality following hip fracture and to increase the likelihood of discharge from hospital. In 2018, 20% of patients failed to achieve the early remobilisation target, due to pain and/or hypotension, factors which might have been anticipated by clear perioperative protocols and closer working between surgery and anaesthetic colleagues.

Current AAGBI guidelines describe core principles of the peri-operative management of people with hip fracture, with one of their aims recommending a peripheral nerve block immediately prior to operative fixation of a hip fracture (in the Emergency Department and at the time of surgery, provided six hours have passed between blocks). There are two peripheral nerve blocks commonly used in the perioperative setting of hip fracture repair, namely femoral or fascia iliaca block. Both techniques have been proven to be safe and efficacious, however, these peripheral nerve blocks have been associated with some residual muscle weakness and increased falls risk which further hampens the ability of a patient to remobilize post-operatively. There is a clinical need to establish a safe, reliable regional anaesthetic technique that will still offer long-acting opioid sparing analgesia, yet minimise the associated motor blockade in order to improve and facilitate remobilization. By also potentially interrupting the sympathetically mediated pain in the lower limb following hip surgery through the blockade of this lumbar sympathetic plexus, it may provide an avenue to produce significant analgesia without causing somatic sensory deficits (e.g. residual motor weakness), thereby facilitating early remobilisation and enhanced recovery. This is not a new technique, rather it is a new approach to a very well established and utilized technique (the psoas compartment block) which has been shown to be very effective, this approach is expected to be as efficacious and potentially safer than previous approaches as it avoids the nerve roots. In terms of the side effect profile of this novel approach to the PCB - there are no new expected side effects above the standard previously explained effects that can occur with any regional technique (for example, haematoma/ LAST / Neuropraxia). This approach would theoretically be associated with a lower side effect profile than previous landmark or current ultrasound-guided PCB technique as it avoids the risk profile of traversing the psoas muscle body and near the exit of the lumbar plexus nerve roots.

This study aims to follow up on the inital case series discussed above to evaluate the efficacy of the SPF block for post op analgesia in patients undergoing hemiarthroplasty surgery.

Aims and Objectives:

This will be a randomised control trial. The primary aim of this study is to further evaluate the efficacy of a sub-psoas muscle fascial plane regional block for providing adequate opioid-sparing/reducing post-operative analgesia, in comparrisson to patients who do not receive a regional anaesthesia block and standard analgesic regieme.

The secondary aim of this study is to explore patients' experience post-operatively in terms of their pain, time to remobilisation, total analgesic requirements, and quality of recovery.

Study End Points/Primary Objectives:

* To evaluate the post-operative analgesia provided by the proposed regional anaesthesia block, utilising:
* Quality of Recovery 15 (QoR15) Score
* Pain scores (Numerical rating scales, Pain Map, VAS, NRS)
* Intraoperative and Postoperative Opioid Requirements Quantification
* Time to remobilisation post-operatively
* (see supplementary material)

Study Design:

This trial will take place in the Anaesthetic and Orthopaedic Departments, University Hospital Galway. All participants will be treated with either the sub-psoas fascial plane block pre or post-operatively, or no regional anaesethesia with a standard analgesic regieme. written consent will be obtained from each participant. Where informed consent is attained, a clinical note review will take place in addition to the psoas muscle sympathetic chain block pre-operatively. Patients will be closely monitored throughout the procedure and surgery. They will be followed up in the post-anaesthetic care recovery unit to assess their pain, in addition to on day one and two on the ward where a full assessment of their recovery, pain, opioid requirements and overall post-operative course will be carried out by the anaesthetic team member involved in this study.

Study Methodology:

In this RCT, all patients enrolled will be undergoing either emergency hip surgery under the orthopaedic team in the theatre complex in University Hospital Galway. Ethical approval from the Galway Clinical Research Ethics Committee will be sought. Once approved, the procedure will be explained at length by the primary research or co-investigators to the patient and all questions will be addressed. The aim would be to provide a timeframe for the patient to consider the procedure before providing consent (i.e. during pre-operative assessment on the ward the night before or morning of their surgery and undergoing the consent process when in the theatre complex). If the patient is agreeable, verbal informed consent will be obtained. a clinical note review will take place to attain basic demographic and clinical data including diagnosis, indication for surgery, type of surgery, type of anaesthetic technique, comorbidities, preadmission opioid requirements. The procedure will be explained at length to the patient and if agreeable to proceed, the patient will be monitored closely as normally would occur in the theatre setting, they will be positioned in theatre briefly onto their lateral side. Under ultrasound-guidance the regional nerve block will be performed by the experienced consultant anaesthesiologist, whereby 30ml of 0.75% Ropivicaine will be slowly injected into the subpsoas fascial plane, whilst at all times throughout and following the procedures the patient will be closely haemodynamically monitored. The patient will be followed up in the recovery post-anaesthetic care unit up to four hours following their surgery. They will then be reviewed by the one of the co-investigators at a timeframe of 0-24 hours and 24-48 hours post-operatively to further establish their analgesic efficacy, their pain scores (see supplementary appendix), quality of recovery, time to remobilization and opioids requirements, ensuring the patient is comfortable and aiming to maximize their recovery period.

This is not a new technique, rather it is a new approach to a very well established and utilized technique - the psoas compartment block (PCB). The PCB utilizes a posterior approach whereby it traverses through the body of the psoas muscle thereby carrying the small risk profile of being near the plane of where the lumbar plexus roots exit the body of the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing orthopaedic surgery at the hip joint in University College Hospital, Galway.
* Individuals over 18 years of age.
* Individuals treated with psoas muscle sympathetic nerve blocks as part of multi-modal analgesic management.
* Individuals with the capacity to make an informed decision regarding study participation.
* Patients that provide written and verbal informed consent.
* Patients whom have not received a fascia iliacus block in the emergency department prior to their surgery.

Exclusion Criteria:

* To be eligible, a patient must have none of these exclusion criteria
* Individuals unable to provide informed consent.
* Individuals < 18 years of age.
* Individuals with an intellectual disability (IQ < 70), cognitive impairment, delirium or with dementia.
* Allergy to the local anaesthesia block components.
* Patients with absolute or relative contraindication to peripheral nerve blocks.
* Coagulopathy (Prothrombin time/International Normalized Ratio of more than 1.50, Activated Partial Thromboplastin Time of more than 60 seconds).
* Cases judged to be inappropriate by the chief investigator.
* Patients whom have received a fascia iliacus block in the emergency department prior to their surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients enrolled will be undergoing Emergency HemiArthroplasty in the theatre complex in University Hospital Galway.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-13 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Efficacy of SPF Block - Quality of Recovery | 48 hours
  Quality of Recovery 15 (QoR15) Score
  a patient-reported outcome measurement measuring QoR after surgery and anesthesia.
  minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).
Opioid Consumption | 48 hours
  Intraoperative and Postoperative Opioid Requirements Quantification
Pain Score | 48 hours
  Pain score - NRS - Numerical Rating Score
  requires the patient to rate their pain on a defined scale. 0-10 where 0 is no pain and 10 is the worst pain imaginable

SECONDARY OUTCOMES:
Time to remobilisation post-operatively | 48hrs
  Time to remobilisation post-operatively